CLINICAL TRIAL: NCT05819138
Title: Type 1 Diabetes Impacts of Semaglutide on Cardiovascular Outcomes
Acronym: T1-DISCO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0794; R01HL165433 (NIH)
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive 0.25 mg once weekly semaglutide injection for 4 weeks.
  Participants will receive 0.50 mg once weekly semaglutide injection for 4 weeks.
  Participants will receive 1.0 mg once weekly semaglutide injection for 6 months.
  Interventions: Drug: Semaglutide Pen Injector
- Placebo (Placebo Comparator): Participants will receive 0.25 mg once weekly placebo injection for 4 weeks. Participants will receive 0.50 mg once weekly placebo injection for 4 weeks. Participants will receive 1.0 mg once weekly placebo injection for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Semaglutide injection
  Other Names: Ozempic
  Arms: Semaglutide
Drug: Placebo — Semaglutide placebo injection
  Arms: Placebo

SUMMARY:
This trial plans to learn more about the effects of a medication, semaglutide, on cardiovascular function, kidney function, and insulin sensitivity in adults with type 1 diabetes. This medication has been effective in reducing cardiovascular disease and diabetic kidney disease and improving glucose control and BMI in adults with type 2 diabetes. This study aims to look at how well the medication works in people with type 1 diabetes. Semaglutide is not approved by the FDA to be used in this way. These procedures are considered to be experimental.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years
* 1) T1D diagnosis defined as positive T1D-associated antibody(ies) or 2) a clinical diagnosis of T1D plus insulin requirement since diagnosis
* Insulin pump or automated insulin delivery systems
* Estimated glomerular filtration rate (eGFR) ≥ 45 ml/min/1.73m2
* Stable doses of drugs altering cardiovascular and renal function (e.g., Angiotensin-Converting Enzyme Inhibitor (ACEi), Angiotensin Receptor Blocker (ARB), statins, diuretics)
* BMI 20-45 kg/m2
* Adequate contraceptive method for females

Exclusion Criteria:

* HbA1c >9%, recent diabetic ketoacidosis (DKA) or hospitalization
* Major congenital heart disease, anemia, severe non-proliferative retinopathy, proliferative retinopathy
* History/family history of medullary thyroid carcinoma, multiple endocrine neoplasia type 2 (MEN2), pancreatitis
* Current/planned pregnancy or nursing
* Uncontrolled thyroid disease or hypertension (HTN) (≥ 160/100 mm Hg despite optimal therapy)
* Use of other non-insulin diabetes medications, insulin sensitizing medications, or systemic steroids in past 3 months
* Use of atypical antipsychotics
* Significant systemic illness such as cancer
* Shellfish/iodine allergy (only exclusionary to iohexol clearance procedure)
* MRI or PAH contraindications (only exclusionary to MRI and PAH procedures), GLP-1RA allergy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Ascending Aortic Pulse Wave Velocity (AA PWV) | Baseline, month 8
  AA PWV is a measure of central arterial stiffness. A lower value indicates a better outcome.
Change in Carotid and Femoral Artery Pulse Wave Velocity (CF-PWV) | Baseline, month 8
  CF-PWV is a measure of peripheral arterial stiffness. A lower value indicates a better outcome.
Change in Carotid and Radial Artery Pulse Wave Velocity (CR-PWV) | Baseline, month 8
  CR-PWV is a measure of peripheral arterial stiffness. A lower value indicates a better outcome.

SECONDARY OUTCOMES:
Change in Insulin Sensitivity | Baseline, month 8
  Insulin Sensitivity is a measure of how well the body responds insulin. A higher value indicates a better outcome; a lower value indicates a worse outcome.
Change in Renal Vascular Resistance (RVR) | Baseline, month 8
  RVR is a measure of mean arterial pressure to renal blood flow. A higher value indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Petter M Bjornstad, MD, Principal Investigator — University of Colorado, Denver; Kristen Nadeau, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Washington Medicine Diabetes Institute (UWMDI), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No